CLINICAL TRIAL: NCT03230227
Title: Presternal Local Analgesia for Postoperative Pain Relief After Open Heart Surgery
Brief Title: Presternal Magnesium With Bupivacain Versus Bupivacain Only for Postoperative Pain Relief in Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00009912
Record Dates: First submitted 2017-07-14; First posted 2017-07-26 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: post open heart surgery pain alleviation
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine magnesium (Active Comparator): ( bupivacain 0.125% magnesium sulfate 5%) infusion in the presternum , for 48 hours
  Interventions: Drug: Bupivacaine magnesium
- bupivacain only (Active Comparator): bupivacaine 0.125% infusion in the presternum , for 48 hours
  Interventions: Drug: Bupivacaine only

INTERVENTIONS:
Drug: Bupivacaine magnesium — bupivacain 0.125% magnesium sulfate 5%) infusion in the presternum , for 48 hours
  Arms: Bupivacaine magnesium
Drug: Bupivacaine only — bupivacaine 0.125% infusion in the presternum , for 48 hours
  Arms: bupivacain only

SUMMARY:
Effective pain relief after cardiac surgery has assumed importance with the introduction of fast track discharge protocols that requires early weaning from mechanical ventilation. Inadequate pain control reduces the capacity to cough, mobility, increases the frequency of atelectasis, and prolongs recovery. Infiltration of local anesthetics near the surgical wound has shown to improve early postoperative pain in various surgical procedures.

Magnesium is the fourth most plentiful cation in our body. It has antinociceptive effects in animal and human models of pain.

DETAILED DESCRIPTION:
Effective pain relief after cardiac surgery has assumed importance with the introduction of fast track discharge protocols that requires early weaning from mechanical ventilation. Inadequate pain control reduces the capacity to cough, mobility, increases the frequency of atelectasis, and prolongs recovery.

A major cause of pain after cardiac surgery is the median sternotomy particularly on the first two postoperative days.

The most often used analgesics in these patients are parenteral opioids which can lead to undesirable side-effects as sedation, respiratory depression, nausea, and vomiting.

Infiltration of local anesthetics near the surgical wound has shown to improve early postoperative pain in various surgical procedures.

Magnesium is the fourth most plentiful cation in our body. It has antinociceptive effects in animal and human models of pain.

It has been mentioned in a systematic review that it may be worthwhile to further study the role of supplemental magnesium in providing perioperative analgesia, because this is a relatively harmless molecule, is not expensive and also because the biological basis for its potential antinociceptive effect is promising.

These effects are primarily based on physiological calcium antagonism, that is voltage-dependent regulation of calcium influx into the cell, and noncompetitive antagonism of N-methyl-D-aspartate (NMDA) receptors.

there is a need to evaluate and compare local magnesium with bupivacaine , in comparison to bupivacain

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* American Society of Anesthesiologists physical status II and III
* Patients scheduled for open heart surgery with sternotomy

Exclusion Criteria:

* - Emergency surgery
* Clinically significant kidney or liver disease
* Patients allergic to local anesthetic
* Patients with prolonged CPB time (>120 min)
* Patients required intra-aortic balloon pump

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 2 days
  assessing VAS scale

SECONDARY OUTCOMES:
hemodynamics | 24 hours
  mean arterial blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided